CLINICAL TRIAL: NCT06568653
Title: The Efficacy of Human Placenta Mesenchymal Stem Cells Derived Exosomes Injection for Treatment of Complex Anal Fistula in Colorectal Surgery Department of Imam Khomeini Hospital Complex: A Non-randomized Clinical Trial.
Brief Title: Human Placenta Mesenchymal Stem Cells Derived Exosomes Injection for Treatment of Complex Anal Fistula
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IR.TUMS.IKHC.REC.1403.113
Record Dates: First submitted 2024-07-22; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-07

CONDITIONS: Fistula Perianal
Keywords: fistula, perianal fistula, non-Crohn's disease, exosome, mesenchymal stem cell, human placenta stem cell
MeSH Terms: conditions — Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention (Experimental)
  Interventions: Procedure: exosome
- control (Active Comparator)
  Interventions: Procedure: routine conventional fistulotomy

INTERVENTIONS:
Procedure: exosome — human placenta mesenchymal stem cell-derived exosome
  Arms: intervention
Procedure: routine conventional fistulotomy — routine conventional fistulotomy
  Arms: control

SUMMARY:
The goal of this clinical trial is to learn if human placenta mesenchymal stem cells (MSC)-derived exosomes work to treat complex perianal fistula in adults without Crohn's disease. The safety of this treatment will also be learned. The main questions it aims to answer are:

* Does treatment with MSC-derived exosomes lower the number of fistula recurrences in participants?
* Is treatment with MSC-derived exosomes safe? We will compare treatment with MSC-derived exosomes to the routine treatment which is fistulotomy (surgery to close the fistula) alone to see if MSC-derived exosomes work better to treat complex fistula.

Participants will:

* Undergo fistulotomy plus MSC-derived exosome injections or fistulotomy alone.
* Visit the clinic the week after surgery and then every 4 weeks for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

* participants with complex perianal fistula
* provided written informed consent

Exclusion Criteria:

* participants with any inflammatory bowel diseases
* pregnant or lactating participants
* participants with contraindications for surgery
* participants with hepatitis
* participants with uncontrolled diabetes
* participants with alcohol or substance abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2024-11-15 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
The number of fistula openings (orifices) will be assessed before and after our intervention. | 3 months
  clinical improvement

SECONDARY OUTCOMES:
QoL questionnaire | 3 months
  quality of life improvement (before and after intervention) assessed by Persian (Farsi) version of the QoLAF (quality of life in patients with anal fistula) questionnaire